CLINICAL TRIAL: NCT04110002
Title: An Injury Prevention Program for Professional Ballet: a Randomized Controlled Investigation
Brief Title: An Injury Prevention Program for Professional Ballet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Joshua D Harris, MD, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00014833
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Accidents Sports; Injury Prevention
Keywords: injury prevention program; professional ballet

STUDY DESIGN:
Intervention Model Description: 2 arm: randomized to injury prevention protocol or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Injury Prevention Program (Experimental): Those allocated to the injury prevention program will be instructed on the program, the added exercises, and the additional time commitment.
  Interventions: Behavioral: Injury Prevention Program
- Control (No Intervention): The control group will practice and perform with no change to pre-existing years' standard operating practice.

INTERVENTIONS:
Behavioral: Injury Prevention Program
  Arms: Injury Prevention Program

SUMMARY:
The aim of this study is to evaluate the efficacy of an injury prevention program for professional ballet dancers.

ELIGIBILITY:
Inclusion Criteria:

* Professional Ballet Dancer
* Willing to participate and undergo informed consent process

Exclusion Criteria:

* Pregnant Women, non-English speaking subjects, or those who decline participation in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-07-15 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Rate of Injury | 1 year
  Number of injuries sustained and reported per subject during the 1 year study. Data will be aggregated according to arm of study to ascertain the rate of injury for each group.

SECONDARY OUTCOMES:
Turn-out degrees | 1 year
  Turn-out degree values to measure flexibility and strength. Turnout is the sum of hip rotation, tibial torsion, and contributions from the foot.
Beighton | 1 year
  Beighton scale to ascertain generalized joint laxity. Maximum score of 9, minimum score of 0.
AOFAS ankle-hindfoot | 1 year
  American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Score. 100 point total score. Instrument combines functional outcome and pain for subject's ankle or hindfoot.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua D Harris, MD, Principal Investigator — The Methodist Hospital Research Institute

IPD SHARING:
Plan to Share IPD: No
Due to privacy concerns, no individual participant data will be available. Only aggregate data may be provided.

REFERENCES:
- [Derived] Vera AM, Barrera BD, Peterson LE, Yetter TR, Dong D, Delgado DA, McCulloch PC, Varner KE, Harris JD. An Injury Prevention Program for Professional Ballet: A Randomized Controlled Investigation. Orthop J Sports Med. 2020 Jul 28;8(7):2325967120937643. doi: 10.1177/2325967120937643. eCollection 2020 Jul. PMID 32782904